CLINICAL TRIAL: NCT05691088
Title: To Evaluate the Clinical Efficacy of Standardized Use of Acetaminophen in Mechanical Ventilation in Children With New Coronary Pneumonia
Brief Title: Clinical Efficacy of Acetaminophen in Mechanical Ventilation in Children With New Coronary Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Clinical Medical College of Jinan University (Other)
Collaborators: Kunming Children's Hospital (Other); Shenzhen Windo Medical Technology Limited Company (Unknown)
Responsible Party: Principal Investigator, Hu Anmin, The Second Clinical Medical College of Jinan University, The Second Clinical Medical College of Jinan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: wm2022001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Acetaminophen,Mechanical Ventilation,Critically Ill Children

STUDY DESIGN:
Intervention Model Description: Clinical efficacy of acetaminophen in mechanical ventilation in children with new coronary pneumonia
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Paracetamol injection
  Interventions: Device: Paracetamol injection
- Group B (No Intervention): Equivalent physiological saline

INTERVENTIONS:
Device: Paracetamol injection — Patients were randomized to receive either paracetamol during mechanical ventilation. When patients were randomized to receive paracetamol (40 mg/kg per day in 4 doses), a placebo infusion of normal saline was administered continuously at the same rate as an equivalent infusion. Placebos could not be distinguished from the active study drug in color, odor, or viscosity.
  In both study groups, IMV was maintained with sufentanil (0-0.2 mcg/kg/h), propofol (0-4 mg/kg/h), and dexmedetomidine (0-1 mcg/kg/h). Assessment of sedation levels by the bedside nurse using the FLACC pain scale to determine if the child is adequately comfortable or in need of more or less medication to maintain adequate ventilation. Assessment of sedation levels by the bedside nurse using the FLACC pain scale (every 6 hours as a minimum time interval).
  Arms: Group A

SUMMARY:
Patients were randomized to receive either paracetamol during mechanical ventilation. When patients were randomized to receive paracetamol (40 mg/kg per day in 4 doses), a placebo infusion of normal saline was administered continuously at the same rate as an equivalent infusion. Placebos could not be distinguished from the active study drug in color, odor, or viscosity.

In both study groups, IMV was maintained with sufentanil (0-0.2 mcg/kg/h), propofol (0-4 mg/kg/h), and dexmedetomidine (0-1 mcg/kg/h). Assessment of sedation levels by the bedside nurse using the FLACC pain scale to determine if the child is adequately comfortable or in need of more or less medication to maintain adequate ventilation. Assessment of sedation levels by the bedside nurse using the FLACC pain scale (every 6 hours as a minimum time interval).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were body weight greater than 1500 g; and mechanically ventilated patients with confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

Exclusion Criteria:

* Exclusion criteria were admitted with a tracheostomy in situ; extracorporeal membrane oxygenation treatment; neurologic dysfunction, hepatic dysfunction, or renal insufficiency; known allergy to or intolerance for paracetamol; and administration of paracetamol in the 24 hours prior to mechanical ventilation.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time | an average of 5 days

SECONDARY OUTCOMES:
Length of ICU stay time | an average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Windo Medical, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No